CLINICAL TRIAL: NCT04118101
Title: Erector Spinae Plane Block for Patients Undergoing Open Renal Surgery Through Flank Incision: A Randomized Controlled Study.
Brief Title: Erector Spinae Plane Block
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Anesthesia and Intensive care clinical researcher, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBRI 2
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: After skin sterilization and draping, a high-frequency linear array ultrasound probe will be placed on the back in a transversly to identify the tip of the T7 transverse process. The tip of the transverse process will be centered on the ultrasound screen and the probe will be rotated into a longitudinally to produce a para-sagittal view, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius and erector spinae muscle. An echogenic 22-G block needle will be inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T7 transverse process. Correct location oft he needle tip in the fascial plane deep to erector spinae muscle will confirmed by injecting 0.5-1 ml normal saline and seeing the fluid lifting the erector spinae muscle off the transverse process without distending the muscle.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Active Comparator): A total of 25 ml bupivacaine 0.5% willbe injected into the ESP.
  Interventions: Drug: ESPB block
- Control group (Placebo Comparator): The ESPB will not be performed.
  Interventions: Other: control

INTERVENTIONS:
Drug: ESPB block — A total of 25 ml bupivacaine 0.5% will be injected into the ESP.
  Arms: ESPB group
Other: control — no ESPB will be given.
  Arms: Control group

SUMMARY:
Erector spinae plane block (ESPB) is a relatively new plane block that was first described by Forero et al. in 2016, to manage persistent neuropathic pain following malunited rib fracture and persistent post-thoracotomy neuropathic pain.It's a relatively simple, ultrasound guided block in which the local anesthetic drugs are injected in the plane between the erector spinae muscle and the vertebral transverse process.This allows the injected local anesthetics to block the ventral and dorsal rami of the spinal nerves in the paravertebral area.

The literature reveals successful case reports denoting the use of ESPB for pain control in cases of acute kidney transplant,percutaneous nephrolithomy, abdominal surgeries including laparoscopic and open nephrectomy, and nephrectomy in the pediatric population.

The aim of this prospective randomized controlled study is to investigate the efficacy of ESPB for pain control in adult patients undergoing open renal surgery through a flank incision with respect to pain scores, postoperative analgesia consumption and patient satisfaction.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study which will be conducted in the Anesthesiology Department at Theodor Bilharz Research Institute after approval by the institutional review board and obtaining patient informed consent. 46 patients will be enrolled in the study and will be randomized to be equally divided into two groups: ESPB group(E group) and control group (C group).

Anesthetic technique:

A preoperative assessment, including a history, physical examination, review of laboratory data, and assignment of ASA classification will be performed on all patients prior to the procedure. After premedication with intravenous midazolam 2 mg, patients will be transferred to the operating room.

Standard monitors such as noninvasive blood pressure, electrocardiography (ECG), and pulse oximetry (SpO2) will be attached. Anesthesia will be induced using propofol 1-2 mg/kg, fentanyl 1-2 µg/kg and sevoflurane. After adequate manual ventilation, atracurium 0.5 mg/kg will be administered to facilitate endotracheal intubation. Ventilation will be started with oxygen and medical air (FiO2 = 0.6). Patients will be positioned in the lateral position to perform the ESPB and for preparation for surgery.

Erector SpinaePlane Block technique:

After skin sterilization and draping, a high-frequency linear array ultrasound probe will be placed on the back in a transverse orientation to identify the tip of the T7 transverse process. The tip of the transverse process will be centered on the ultrasound screen and the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius and erector spinae muscle.The rhomboid major muscle has its lower border a tthe T5-6 vertebral level and its absence will be used as additional confirmation that the T7 transverse process is being viewed. An echogenic 22-G block needle will be inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T7 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle will confirmed by injecting 0.5-1 ml normal saline and seeing the fluid lifting the erector spinae muscle off the transverse process without distending the muscle.

ESPB group:

A total of 25 ml bupivacaine 0.5% will be injected into the ESP.

Control group:

The ESPB will not be performed. Surgical technique and postoperative care will follow standard local clinical practice.

Pain management:

Numerical Rating Scale (NRS) pain score will be used immediately postoperatively and then at 30 minutes, 1, 2, 4, 6, 12 and 24 h. Scores (1-3) are considered mild pain, (4-6) moderate pain and (7-10) severe pain. Rescue analgesia with intravenous pethidine (25 mg) will be prescribed if the patient's resting NRS score is more than three or on patient demand. Additional intravenous doses of 25 mg of pethidine will be given if needed to achieve a score below 4. The second rescue analgesic plan will be intravenous ketorolac 30 mg diluted in 100 ml normal saline and administered slowly, if NRS remained persistently >3 after 15 min of the first rescue analgesic administration.

Data collection

1. Age
2. Sex
3. BMI
4. ASA Classification
5. Intraoperative and postoperative arterial blood pressure
6. Intraoperative and postoperativeheart rate
7. Numerical Rating Scale (NRS) pain score immediately postoperatively and then at 30 minutes, 1, 2, 4, 6, 12 and 24 h.
8. Postoperative analgesia consumption
9. The overall degree of patient satisfaction will be assessed using a three-point scale (good, moderate, and bad) on the first postoperative day.
10. Block related complications (e.g Pneumothorax)
11. Postoperative opioid related complications (e.g. Nausea, vomiting, constipation, sedation)

Statistics:

The patients will be randomly divided into two groups; group (E) and group (C). Forty-six patients will be prospectively enrolled for each study of patients who had been diagnosed to be able to reject the null hypothesis that the population means of the groups are equal with Power calculations suggested that a minimum of 23 subjects per group will be required to detect 10% difference in time for first rescue analgesia between groups (taking type I or α error of 5%, type II or β error of 20% and Standard Deviation=10). To be on a safer side, patients will be included in each group (n=23).

Statistical analyses will be performed using JMP ver. 12.0 (SAS Institute Inc., Cary, NC, USA). The number of patients who will be reported complications corresponding percentage (%) for nominal variables; for continuous variables with normal distribution, and the Mann-Whitney U test will be used for nonparametric variables. The level of significance for both the tests set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide a written informed consent.
* ASA I-II.
* Patient is scheduled to perform an elective open renal surgery through a flank incision.

Exclusion Criteria:

* ASA III-IV
* Pregnancy.
* Patient is allergic to bupivacaine local anesthetic.
* Impaired coagulation (Platelet count< 150,000 cells/mcl and/or INR ≥ 1.4).
* Infection at site of injection.
* Prior same side flank surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 30-45 minutes.
  Rescue analgesia with intravenous pethidine (25 mg) will be prescribed if the patient's resting NRS score is more than three or on patient demand. Additional intravenous doses of 25 mg of pethidine will be given if needed to achieve a score below 4. The second rescue analgesic plan will be intravenous ketorolac 30 mg diluted in 100 ml normal saline and administered slowly, if NRS remained persistently >3 after 15 min of the first rescue analgesic administration.

SECONDARY OUTCOMES:
Postoperative analgesic consumption | over the first 24 hours post operatively.
  amount of total analgesics required post operatively.
Patient satisfaction | over first 24 hours post operatively.
  measuring degree of patient discomfort and amount of analgesics required.

CONTACTS AND LOCATIONS:
Overall Officials: Moshira S Mohamed, MD, Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available as excel sheets supplemented with the results but other personal data won't be available to ensure patient privacy.
Supporting Information: Study Protocol
Time Frame: 1 year

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016